CLINICAL TRIAL: NCT05515848
Title: Regional, Multicentric Registry of Aortic Valve-sparing Root Replacement, According to the Inclusion Technique Described by Tirone David
Brief Title: Aortic Valve-sparing Root Replacement, According to the Inclusion Technique Described by Tirone David
Acronym: AORTLANTIC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0540
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Aortic Root Aneurysm; Aortic Regurgitation
Keywords: Valve-sparing aortic root replacement; David procedure; Acute aortic dissection; Aortic Regurgitation; Bicuspid aortic valve; French multicentric registry
MeSH Terms: conditions — Aortic Root Aneurysm; Aortic Valve Insufficiency; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AORTLANTIC registry: Patients undergoing aortic root surgery with aortic valve conservation, using the inclusion technique described by Tirone David, between January 1, 2004 and December 31, 2021, at five centers (Nantes - Rennes - Brest - Angers - Tours University Hospital (UH))
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this retrospective study.

SUMMARY:
Retrospective observational study of all patients undergoing aortic root surgery with aortic valve conservation, using the inclusion technique described by Tirone David, between January 1, 2004 and December 31, 2020, at six centers (Nantes - Rennes - Brest - Angers - Tours [two centers]). The main objective of this study is to evaluate the survival without re-intervention for aortic valve dysfunction (surgery or TAVI).

DETAILED DESCRIPTION:
Retrospective observational study of all patients undergoing aortic root surgery with aortic valve conservation, using the inclusion technique described by Tirone David.

Inclusion criteria: Patients undergoing aortic root surgery with conservation of the aortic valve, according to the inclusion technique described by Tirone David, between January 1, 2004 and December 31, 2020, at one of the six centers: Nantes, Rennes, Brest, Angers, Tours (two centers).

Non-inclusion criteria: Prosthetic replacement of the aortic valve intraoperatively during the first operation.

Objectives and endpoints :

* The survival without re-intervention for aortic valve dysfunction (surgery or TAVI)
* The overall cardiovascular survival
* The survival without aortic insufficiency of grade equal to or greater than two
* The survival without aortic infective endocarditis
* Assessment of long-term stroke risk Assessment of the risk of a major bleeding event in the long term Data analysis : The AORTLANTIC study is included in the EPICARD registry which is the official, national database of the French Society of Cardiac Surgery. Study data will then be collected using EPICARD's electronic Case Report Form (eCRF) and then analyzed using a multivariate Cox model. For the follow-up, the WEPI eCRF is used.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing aortic root surgery with conservation of the aortic valve, according to the inclusion technique described by Tirone David, between January 1, 2004 and December 31, 2021, at one of the six centers: Nantes, Rennes, Brest, Angers,Tours UH.

Non inclusion criteria :

* Prosthetic replacement of the aortic valve intraoperatively during the first operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing aortic root surgery with aortic valve conservation, using the inclusion technique described by Tirone David, between January 1, 2004 and December 31, 2021, at five centers (Nantes, Rennes, Brest, Angers,Tours UH) .
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2021-11-07 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the survival without re-intervention for aortic valve dysfunction (surgery or TAVI), after aortic root surgery with conservation of the aortic valve, according to the inclusion technique described by Tirone David | Conditional survival starting at 30 days
  Number of patients alive without re-intervention for aortic valve dysfunction (surgery or TAVI)

SECONDARY OUTCOMES:
Evaluate the overall cardiovascular survival results | up to 17 months
  Number of patients alive
Evaluate the absence of aortic insufficiency greater than or equal to grade two between the two types of aortic tube graft (right prosthesis or Valsalva prosthesis) | up to 17 months
  Number of patients alive without aortic insufficiency of grade equal to or greater than two
Evaluate the risk of infective endocarditis | up to 17 months
  Number of patients alive without aortic infective endocarditis
Evaluate the risk of stroke | up to 17 months
  Number of patients alive without stroke
Evaluate the risk of major bleeding event | up to 17 months
  Number of patients alive major bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christian ROUSSEL, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No